CLINICAL TRIAL: NCT00599755
Title: A Multicenter Phase Ib Trial to Measure [18F]-Fluorodeoxyglucose Uptake by Positron Emission Tomography in Stage IIIB and IV Non-Small Cell Lung Cancer Before and After Chemotherapy With Gemcitabine and Cisplatin or Carboplatin
Brief Title: Phase I Imaging Study Evaluating Gem/Cis or Gem/Carbo for Participants With Non-Small Cell Lung Cancer (MK-0000-083 AM3)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0000-083; 2007_662 (Other: Merck)
Record Dates: First submitted 2008-01-07; First posted 2008-01-24 (Estimated); Results first posted 2012-06-27 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Carcinoma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gem/Cis or Gem/Carbo (Experimental)
  Interventions: Radiation: Comparator: CT or MRI and FDG-PET; Drug: Gemcitabine and Cisplatin or Gemcitabine and Carboplatin

INTERVENTIONS:
Radiation: Comparator: CT or MRI and FDG-PET — Participants have 4 computed tomography (CT) or magnetic resonance imaging (MRI) scans at screening, baseline, at the end of each treatment cycle (day 21 and day 42.) They also have FDG-PET scans, 2 at Baseline and one at the end of each treatment cycle.
Drug: Gemcitabine and Cisplatin or Gemcitabine and Carboplatin — Gemcitabine administered intravenously at a dose of 1000-1250 mg/m^2 on Day 1 and Day 8 of each cycle; Cisplatin administered intravenously at a dose of 60-85 mg/m^2 or Carboplatin at a dose of 4-6 Area Under the Curve (AUC) on Day 1 of each cycle. Two cycles are given 3 weeks apart.

SUMMARY:
This study will use imaging to look at tumor response to combination chemotherapy of gemcitabine (Gem) and cisplatin (Cis) or gemcitabine and carboplatin (Carbo) in non small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytopathologically confirmed metastatic or locally advanced stage IIIB/IV Non-small cell lung cancer (NSCLC)
* Has measurable disease
* Has not been previously treated with surgery (involving the thorax), radiation (unless it was for a metastatic site), or chemotherapy for NSCLC
* Is 18 years of age or older
* Has a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Women of childbearing potential have a negative pregnancy test

Exclusion Criteria:

* Is participating in or has participated in a study with an investigational compound or device within 30 days or 5 half-lives of the start of treatment
* Has untreated brain metastases related to their NSCLC or carcinomatous meningitis
* Abuses drugs or alcohol
* Is pregnant or breastfeeding
* Is Human Immunodeficiency Virus (HIV) positive
* Has active viral hepatitis
* Has hearing loss
* Has poorly controlled diabetes mellitus
* Is allergic to gemcitabine, cisplatin or carboplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2010-06-10 (Actual); Study Completion 2011-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Cisplatin or Gemcitabine and Carboplatin: Tumor uptake of FDG is imaged by PET both before and after combination chemotherapy with Gem/Cis or Gem/Carbo
Period: Overall Study
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Started | 68
Completed | 49
Not Completed | 19
Not completed — Adverse Event | 11
Not completed — Withdrawal by Subject | 2
Not completed — Progression of Disease | 3
Not completed — Other Reason | 2
Not completed — No data available | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Response Conversion Rate Between 3 and 6 Weeks After Starting Chemotherapy at a Threshold of a 20% Decrease in SUVmean
Description: Metabolic response conversion rate is the number of participants initially classified as non-metabolic responders relative to baseline at week 3 after starting chemotherapy, who are then, relative to week 3, reclassified as metabolic responders at week 6 after starting chemotherapy, based on a pre-specified threshold of a 20% decrease in mean standardized uptake value (SUVmean) of [18F]-Fluorodeoxyglucose (FDG). The SUVmean was calculated by summing the radioactivity from volumes of interest within each tumor and normalizing for the injected dose and lean body mass.
Time Frame: Weeks 3 and 6 following chemotherapy
Population: Participants with evaluable scans classified as non-metabolic responders relative to baseline at 3 Weeks after starting chemotherapy
Measure: Number; unit: Participants
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Number analyzed (Participants) | 25
Participants | 10
Statistical Analysis 1: Comparison: Gemcitabine and Cisplatin or Gemcitabine and Carboplatin; Test type: Superiority or Other; Proportion = 0.4, 80% CI 2-sided [0.27 to 0.55]

2. Secondary Outcome: Repeatability of FDG SUVmean at Baseline
Description: Two positron emission tomography (PET) scans are obtained on different days at baseline, as close together as possible, under conditions of no biological change, to measure FDG SUVmean. The SUVmean was calculated by summing the radioactivity from volumes of interest within each tumor and normalizing for the injected dose and lean body mass.
Time Frame: Between -14 to -6 days and between -5 to 0 days prior to starting chemotherapy
Population: Participants who underwent two baseline PET scans
Measure: Geometric Mean (Standard Deviation); unit: SUVmean
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Number analyzed (Participants) | 64
SUVmean | 3.79 (1.14)
Statistical Analysis 1: Comparison: Gemcitabine and Cisplatin or Gemcitabine and Carboplatin; Test type: Superiority or Other; Concordance correlation coefficient = 0.88, 80% CI 2-sided [0.85 to 0.92]

3. Secondary Outcome: Change in FDG-PET Uptake From Baseline to Week 3
Description: Fold change in SUVmean of FDG uptake with accompanying 80% Confidence Interval. The SUVmean was calculated by summing the radioactivity from volumes of interest within each tumor and normalizing for the injected dose and lean body mass.
Time Frame: Baseline and Week 3
Population: Participants with PET scans at baseline and 3 weeks after starting chemotherapy
Measure: Number (90% Confidence Interval); unit: Fold Change in SUVmean
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Number analyzed (Participants) | 54
Fold Change in SUVmean | 0.75 [0.70 to 0.80]

4. Secondary Outcome: Change in FDG-PET Uptake From Week 3 to Week 6
Description: as for outcome 3
Time Frame: Week 3 and Week 6
Population: Participants with PET scans at 3 weeks and 6 weeks after starting chemotherapy
Measure: Number (90% Confidence Interval); unit: Fold change in SUVmean
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Number analyzed (Participants) | 47
Fold change in SUVmean | 0.85 [0.81 to 0.90]

5. Secondary Outcome: Change in FGD-PET Uptake From Baseline to Week 6
Description: as for outcome 3
Time Frame: Baseline and Week 6
Population: Participants with PET scans at baseline and 6 weeks after starting chemotherapy.
Measure: Number (90% Confidence Interval); unit: Fold change in SUVmean
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Number analyzed (Participants) | 47
Fold change in SUVmean | 0.65 [0.60 to 0.71]

6. Post Hoc Outcome: Metabolic Response Conversion Rate Between 3 and 6 Weeks After Starting Chemotherapy At a Threshold of a 30% Decrease in SUVmean
Description: Metabolic response conversion rate is the number of participants initially classified as non-metabolic responders relative to baseline at week 3 after starting chemotherapy, who are then, relative to week 3, reclassified as metabolic responders at week 6 after starting chemotherapy, based on a pre-specified threshold of a 30% decrease in SUVmean of [18F]-Fluorodeoxyglucose (FDG). The SUVmean was calculated by summing the radioactivity from volumes of interest within each tumor and normalizing for the injected dose and lean body mass.
Time Frame: Weeks 3 and 6 following chemotherapy
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Number analyzed (Participants) | 32
Participants | 4
Statistical Analysis 1: Comparison: Gemcitabine and Cisplatin or Gemcitabine and Carboplatin; Test type: Superiority or Other; Proportion = 0.125, 80% CI 2-sided [0.06 to 0.23]

ADVERSE EVENTS:
Arm/Group | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin
Serious Adverse Events (participants affected / at risk) | 24/68
Other Adverse Events (participants affected / at risk) | 61/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Lung abscess (Infections and infestations) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Cisplatin or Gemcitabine and Carboplatin (N=68)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 11 (12)
Constipation (Gastrointestinal disorders) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 28 (29)
Vomiting (Gastrointestinal disorders) | 10 (10)
Asthenia (General disorders) | 7 (7)
Chest pain (General disorders) | 5 (5)
Fatigue (General disorders) | 14 (14)
Pyrexia (General disorders) | 8 (8)
Neutrophil count decreased (Investigations) | 6 (7)
Decreased appetite (Metabolism and nutrition disorders) | 17 (17)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Subsequent to multicenter publication, or 24 months after study completion, whichever comes first, an investigator and/or colleague(s) may publish the results for their study site independently. The SPONSOR recommends against this practice due to scientific concerns. The SPONSOR must have the opportunity to review all publications or presentations regarding this study 60 days prior to submission, and any information identified by the SPONSOR as confidential must be deleted prior to submission.